CLINICAL TRIAL: NCT04160650
Title: Educational Nursing Intervention on Nutrition Impact Side-effects' Self-care Among Patients With Colorectal Cancer During Chemotherapy: A Research Protocol for a Randomised Controlled Trial
Brief Title: Educational Nursing Intervention Among Patients With Colorectal Cancer During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leena Tuominen, Principal Investigator, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NursEff
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Patient Empowerment; Patient Activation; Self Care; Cancer of Colon; Cancer of Rectum
MeSH Terms: conditions — Patient Participation; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A two-arm, single center, patient blinded superiority trial with stratified randomization (1:1) and with repeated measures
Who Masked: Participant
Masking Description: Participants are blinded after assignment to interventions, those in intervention and control groups are not aware which treatment they get.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational nursing intervention (Experimental): Patients in experimental group receive standard care and one-hour educational session. Patients are provided knowledge of
  * healthy diet
  * malnutrition, its prevalence and consequences for patients with CRC undergoing CT
  * side effects impairing nutrition intake during CT treatment.
  * prevention and self-care methods of the side effects Teach-back is used to verify participants' understanding. Empowering effect is confirmed by using active listening and asking patients' individual side effects, self-care strategies and need of additional knowledge in the beginning of the session and supporting patients' self-care methods when they have been applicable and effective. Additional knowledge of each theme is offered. To reinforce the intervention effect patients receive after the first CT a self-monitoring diary including assessment of side effects prevalence and intensity (NRS 0-10) before and after the self-care strategies. They return diaries by the 5th cycle of CT.
  Interventions: Behavioral: Educational nursing intervention on nutrition intake related chemotherapy induced side-effects' self-care among the patients with colorectal cancer
- Standard care (No Intervention): Patients in control group receive standard care, information of
  * general CT induced side effects and their self-care; nausea, diarrhoea, obstipation and sores in the mouth, peripheral neuropathy symptoms, local venous irritation, heart symptoms, mucous and skin irritation
  * side-effects' self-monitoring, fluid intake, medication dose changes, effect of CT
  * weight control
  * taste alteration
  * cold sensitivity
  * variable diet
  * dietary supplements
  * available dietitian services
  They receive a self-monitoring diary, which includes only side effects and their intensity (NRS 0-10).

INTERVENTIONS:
Behavioral: Educational nursing intervention on nutrition intake related chemotherapy induced side-effects' self-care among the patients with colorectal cancer — This is an educational intervention which aims to answer the questions:
  1. In patients with CRC what is the effect of empowering education versus standard education on knowledge level in 4 months follow-up?
  2. In patients with CRC what is the effect of empowering education versus standard education on activation level related to nutrition impact side effects' self-care in 4 months follow-up?
  3. In patients with CRC what is the effect of empowering education versus standard education on malnutrition risk in 4 months follow-up?
  4. In patients with CRC what is the effect of empowering education versus standard education on QoL in 4 months follow-up?
  Arms: Educational nursing intervention

SUMMARY:
The prevalence of malnutrition is common among patients with colorectal cancer. Chemotherapy induced side effects may impact negatively on nutrition intake thus increase the risk of malnutrition and serious complications for patients. Purpose is to test the effect of empowering education on activation and knowledge level among patients with colorectal cancer during the chemotherapy. Secondary outcomes are quality of life and malnutrition.

A two-arm, single center, patient blinded superiority trial with stratified randomization (1:1) and with repeated measures is used to measure the effectiveness of face-to-face education on nutrition intake related chemotherapy induced side-effects' self-care compared to standard care. Eligibility criteria are adult patients diagnosed with colorectal cancer and receiving intra venous chemotherapy treatment. Patients are recruited in one university hospital outpatient clinic in Finland. Experienced oncology nurse delivers the intervention two weeks after the first chemotherapy. Primary outcomes are activation in self-care and knowledge level. Secondary outcomes are quality of life and risk of malnutrition measured at baseline (M0) and after eight (M1) and 16 weeks (M2) after the intervention.

The study will provide knowledge of nurse-led educational intervention on self-care among patients with colorectal cancer. The findings will contribute to patient education and self-care, thus better quality of life.

DETAILED DESCRIPTION:
The prevalence of malnutrition is common among patients with colorectal cancer. Chemotherapy induced side effects (nausea, vomiting, pain, mouth sores, fatigue, diarrhea, constipation, distress) may impact negatively on nutrition intake thus increase the risk of malnutrition thus serious complications for patients. Nurse-led empowering education may have positive effect on activation and knowledge level and enhance self-care of this patient group. Studies of nurse-led interventions that may enhance nutrition intake are scarce. Therefore, purpose of this study is to test the effect of educational nursing intervention on activation and knowledge level among patients with colorectal cancer during the chemotherapy. Secondary outcomes are quality of life and risk of malnutrition.

A two-arm, single center, patient blinded superiority trial with stratified randomization (1:1) and with repeated measures is used to measure the effectiveness of face-to-face education on nutrition intake related chemotherapy induced side-effects' self-care compared to standard care. Eligibility criteria are adult patients diagnosed with colorectal cancer and receiving intra venous chemotherapy treatment. Patients are recruited in one university hospital outpatient clinic in Finland. Experienced oncology nurse delivers the intervention two weeks after the first chemotherapy. Primary outcomes are activation in self-care and knowledge level. Secondary outcomes are quality of life and malnutrition risk measured at baseline (M0) and after eight (M1) and 16 weeks (M2) after the intervention.

The study will provide knowledge of the effectiveness of nurse-led empowering educational intervention on self-care related to chemotherapy-induced side effects that may deteriorate nutrition intake among patients with colorectal cancer. The findings will contribute to patient education and self-care, thus better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* able to speak and understand Finnish
* receiving chemotherapy every three weeks in outpatient clinic: oxaliplatin+capecitabine= Xelox; irinotecan + capecitabine = Xeliri; Xelox or Xeliri + Bevacizumab

Exclusion Criteria:

* weak physical, psychological or cognitive function that prevents participation
* not able to understand Finnish

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
The rate of knowledge level (Knowledge test of malnutrition, nutrition impact side effects and their self-care, RasOma, Tuominen et al. 2019) | From the baseline to 8 and 16 weeks after the intervention
  Knowledge is seen as essential for empowerment (Rankinen et al. 2014; Castro et al. 2016). It is assumed that knowledge level is better in the intervention group compared to control group. Knowledge test was developed in the research group, which included an oncologist, a dietitian, oncology nurses and a researcher. The instrument includes 15 items (yes/no, right answer=1 point, wrong answer=0 points).
The rate of self care activation (Patient Activation Measure PAM, Insignia Health; Hibbard et al. 2004) | From the baseline to 8 and 16 weeks after the intervention
  Activated individuals have the knowledge, skills and confidence to self-manage their health. PAM shows how ready, willing and able an individual is to manage his or her health and healthcare.It is assumed that patients in the intervention group are more activated to self-care their side effects. The activation score is based on a 0-100 point scale. A change of 3-4 points is associated with the difference between engaging and not engaging in particular behaviors. Activation self care is rated from 1 to 4 (1= low activation level; believing the patient role is important, 2=low activation level; having the confidence and knowledge necessary to take action, 3=moderate activation level; actually taking action to maintain and improve one's health, and 4=high activation level; staying the course even in stressful situations)(InsigniaHealth 2017).

SECONDARY OUTCOMES:
The incidence of malnutrition risk (Nutritional Risk Screening NRS2002, Kondrup et al. 2003) | From the baseline to 8 and 16 weeks after hte intervention
  Nutrition consultations have affected positively on patients' food intake and nutritional status (Kiss & Krishnasamy 2014; Tu et al. 2013; Ravasco 2011, 2012). Patients with a total score of ≥3 are classified as nutritionally at risk. It is assumed that malnutrition risk is lesser in the intervention group compared to control group.
The rate of quality of life (The Functional Assessment of Cancer Therapy Scale - Colorectal, FACT-C, Cella et al. 1993) | From the baseline to 8 and 16 weeks after the intervention
  The risk of malnutrition is strongly associated with QoL in cancer patients initiating chemotherapy (Calderon et al. 2018).The FACT-C questionnaire consists of 36 items on a 5-point Likert scale in four areas of well-being: physical (0-28 points), social (0-28 points), emotional (0-24 points), functional (0-28 points) and CRC subscale (0-28 points). Higher score means better QoL (34 points=low level, 34-68 points= satisfactory, 68-102 points=average and 102-136 points=high)(Ganesh et al. 2016; Goździewicz et al. 2017).

OTHER OUTCOMES:
Incidence of interruption, transfer and cancellation of the treatments | From the baseline to 8 and 16 weeks after the intervention
  Better nutritional status is related to better treatment effect and better well-being, which may lead to better adherence to treatment schedule (Ravasco et al. 2012). Data is collected from patients' records.
Incidence of morbidity | From the baseline to 16 weeks after hte intervention
  Worse nutritional status is related to greater morbidity (Ravasco et al. 2012). Data is collected from patients' records.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Leino-Kilpi, PhD, Principal Investigator — University of Turku
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tuominen L, Ritmala M, Vahlberg T, Makela S, Nikander P, Leino-Kilpi H. The effect of nurse-led empowering education on nutrition impact side effects in patients with colorectal cancer undergoing chemotherapy: A randomised trial. Patient Educ Couns. 2023 Oct;115:107895. doi: 10.1016/j.pec.2023.107895. Epub 2023 Jul 15. PMID 37473602
- [Derived] Tuominen L, Ritmala-Castren M, Nikander P, Makela S, Vahlberg T, Leino-Kilpi H. Empowering patient education on self-care activity among patients with colorectal cancer - a research protocol for a randomised trial. BMC Nurs. 2021 Jun 10;20(1):94. doi: 10.1186/s12912-021-00617-z. PMID 34112154